CLINICAL TRIAL: NCT03963895
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of a Single Dose of E-WE Thrombin, Administered During a Regular Hemodialysis Procedure, in Patients With End-Stage Renal Disease on Chronic Hemodialysis
Brief Title: Safety and Efficacy Study of AB002 (E-WE Thrombin) in End Stage Renal Disease Patients on Chronic Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aronora, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EWE-19-02
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: End Stage Renal Disease; Thrombosis
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AB002 (E-WE-thrombin) Dose 1 (Experimental): Participants will receive a single dose of 1.5 mcg/kg E-WE thrombin.
  Interventions: Drug: AB002 Dose 1
- AB002 (E-WE-thrombin) Dose 2 (Experimental): Participants will receive a single dose of 3.0 mcg/kg E-WE thrombin.
  Interventions: Drug: AB002 Dose 2
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AB002 Dose 1 — AB002 (E-WE thrombin) 1.5 mcg/kg administered on Day 1 as a single intravenous infusion
  Other Names: E-WE thrombin Dose 1
  Arms: AB002 (E-WE-thrombin) Dose 1
Drug: AB002 Dose 2 — AB002 (E-WE thrombin) 3.0 mcg/kg administered on Day 1 as a single intravenous infusion
  Other Names: E-WE thrombin Dose 2
  Arms: AB002 (E-WE-thrombin) Dose 2
Drug: placebo — placebo administered on Day 1 as a single intravenous infusion
  Arms: Placebo

SUMMARY:
This study evaluates the safety and efficacy of AB002 (E-WE thrombin) in patients with end stage renal disease on chronic hemodialysis. Two dose levels will be evaluated in two cohorts. Within each cohort the patients will be randomized to receive either AB002 (E-WE thrombin) or placebo (at a ratio of 2:1 active: placebo).

ELIGIBILITY:
Inclusion Criteria:

1. End Stage Renal Disease (ESRD) maintained on stable outpatient hemodialysis regimen, using an established (> 3 months) and normally functioning, regular flow, uninfected mature AV fistula (or AV graft) and skin consistent with standard chronic hemodialysis access injuries, and hemodialysis stability defined as Kt/V ≥ 1.2 within 3 months prior to screening at a healthcare center for > 3 months from screening.
2. On hemodialysis regimen at least 3 times per week for a minimum of 3 hours per dialysis session, using a complication-free well maintained AV fistula (or AV graft), expected and plan to continue this throughout and for at least 3 months beyond the study.
3. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent and agrees to comply with protocol requirements and study related procedures.
4. Willing to be confined to the clinical research unit for the duration of the study, able to comply with all study-related requirements, and able to adhere to study restrictions and visit schedules.
5. Male or female, between 18 and 80 years of age (inclusive) at the time of screening.
6. Body Mass Index (BMI) of ≥ 18 at the time of screening.
7. Considered by the principle investigator (PI) to be clinically stable with respect to underlying ESRD, based on the medical evaluation that includes medical and surgical history, and a complete physical examination including vital sign measurements, electrocardiograms (ECGs), and clinical laboratory and coagulation test results at screening. Repeat assessments are permitted for any laboratory, coagulation, ECG, or vital sign parameter required for enrollment.
8. Female patients must be of non-childbearing potential and must have undergone one of the following sterilization procedures at least 6 months prior to dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy;

   or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
9. Male patients must either be sterile (vasectomy with history of a negative sperm count following the procedure); practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable); use a male condom with any sexual activity; or agree to use a birth control method considered to be appropriate by the Investigator from the time of dosing until 90 days after study drug administration. Male patients must agree not to donate sperm for a period of 90 days after study drug administration.

Exclusion Criteria:

1. Documented history of acute vasoocclusive thrombotic event (acute coronary syndrome, stroke or transient ischemic attack, venous thromboembolic event), or vascular access fistula or AV graft failure in the past 3 months.
2. With the exception of unfractionated heparin during HD that is allowed until study check-in, concomitant or prior use of anticoagulant/antiplatelet agents (e.g., low molecular weight heparins, warfarin, apixaban, bivalirudin, ticagrelor, edoxaban, dabigatran, rivaroxaban, clopidogrel, prasugrel, ticlopidine, eptifibatide, tirofiban, dipyridamole, diclofenac, and all other non steroidal antiinflammatory drugs) that may affect hemostasis for 2 weeks prior to check in on Day -8 and throughout the study.
3. Any clinically significant (CS) concomitant disease or condition (including treatment for such conditions) that, in the opinion of the PI, could either interfere with the study drug, compromise interpretation of study data, or pose an unacceptable risk to the patient.
4. Any other CS abnormalities in laboratory test results at screening or Day

   * 8 check-in that would, in the opinion of the PI, increase the patient's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
5. Pregnant (positive pregnancy test) at screening or check-in on Day -8. If serum human chorionic gonadotropin (hCG) pregnancy test results are indeterminate, follow-up testing should be performed to determine eligibility. All female patients will not be pregnant and will have a negative pregnancy test at screening and check-in on Day -8, with the following exception: females receiving dialysis with an indeterminate pregnancy test result or persistently low hCG resulting in a false positive pregnancy test may be included in the study at the discretion of the PI. Postmenopausal patients with a result outside the postmenopausal range or an indeterminate pregnancy test will undergo additional testing with FSH to confirm postmenopausal status prior to study enrollment.
6. Treatment with another investigational drug or participation in a device study within 30 days (or 5 half lives, whichever is longer) prior to check-in on Day -8.
7. Acute illness that is considered by the PI to be CS within 2 weeks of check-in on Day 8.
8. Surgery within the past 90 days prior to dosing which in the opinion of the PI or designee is clinically relevant.
9. Currently have established underlying inherited or acquired symptomatic bleeding disorders and/or are at risk for excessive bleeding per PI judgment or current active bleeding (e.g., gastrointestinal, intracranial), aside from minor bleeding from the puncture site on the AV fistula or AV graft, which would be expected to occur during the dialysis procedure, with the following values:

   * Platelet count < 100,000 cells/mm3 (if < 100,000 cells/mm3 but > 75,000 cells/mm3, with permission of PI and medical monitor) at screening or check-in on Day -8.
   * INR > 1.4 at screening or check-in on Day -8
   * aPTT up to 1.2 x upper limit of normal (ULN) (if > 1.2 x ULN and up to < 1.5 x ULN, with permission of PI and medical monitor) at screening or check-in on Day -8
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x ULN at screening or check-in on Day -8
   * Total bilirubin > 1.2 x ULN at screening or check-in on Day -8
   * Hemoglobin concentration < 10 g/dL at screening or check-in on Day

     * 8
10. Seated blood pressure < 90/40 mmHg at screening and check-in on Day

    * 8.
11. Exclusion criteria for ECG at screening and check-in on Day -8:

    Heart rate < 45 and > 110 bpm QTcF interval > 500 msec bpm = beats per minute; msec = milliseconds; QTcF = QT interval corrected using Fridericia's formula
    * Any significant arrhythmia or conduction abnormality, (including but not specific to atrioventricular block [2nd degree or higher], Wolff Parkinson White syndrome [unless curative radio ablation therapy]), which, in the opinion of the PI and Medical Monitor, could interfere with the safety for the individual patient.
    * Non-sustained or sustained ventricular tachycardia (> 2 consecutive ventricular ectopic beats at a rate of > 1.7/second).
12. History of a CS allergy or a known sensitivity or idiosyncratic reaction to any compound known to be present in E-WE thrombin, its related compounds, or any compound listed as being present in the study formulation.
13. Hypersensitivity to ß-lactam / penicillin derivatives.
14. Participate in strenuous exercise from 72 hours prior to check-in on Day -8 and throughout the study.
15. Positive test for drugs of abuse and/or positive alcohol test at screening or check in on Day 8 if not accounted for by a prescription medication. Patients with a positive test based on a prescribed medication may be enrolled.
16. Positive test at screening for hepatitis B surface antigen (HBsAg) or human immunodeficiency virus (HIV). If a patient with ESRD has positive test results for hepatitis C virus (HCV) but liver function tests are otherwise not clinically significant, the patient may be included at the PI's discretion.
17. Receiving blood purification therapy other than HD.
18. Donation of blood or significant blood loss within 56 days prior to dosing.
19. Plasma donation within 7 days prior to dosing.
20. Presence of advanced malignant neoplasms of any organ or system that produces illness or symptoms that have been treated within 3 months with chemotherapy or whole body irradiation, or bone marrow irradiation, and may affect life expectancy in the following 6 months.
21. Any other reason that would render the patient unsuitable for study enrollment at the discretion of the PI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All subject-level clinical, laboratory, samples and imaging data as well as protocols, informed consent forms to participate in the trial, data dictionary, and code book will be preserved for data sharing. Shared data will be deidentifed and all raw data generated in connection with this study will be retained by the Investigator's institution.
  All data will be shared with controlled access. Prior to granting access outside of the Sponsor's archive, data will be deidentified by removing all 18 direct identifiers according to HIPAA Privacy Rule's Safe Harbor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is completed and unblinded, the clinical CRO Celerion will transfer all scientific data to the Sponsor for archival and the Sponsor will update the trial status to "complete" in ClinicalTrials.gov. Data underlying the reported results will be made available 3 months after publication in a peer-reviewed journal for a period of 5 years.
Access Criteria: Potential parties from other organizations can learn about study data and identify whether it could be suitable for their research purposes though summary information (ClinicalTrials.gov, Pubmed) that will be readily available on our website. Data will be made available upon request to Aronora.

REFERENCES:
- [Derived] Verbout NG, Lorentz CU, Markway BD, Wallisch M, Marbury TC, Di Cera E, Shatzel JJ, Gruber A, Tucker EI. Safety and tolerability of the protein C activator AB002 in end-stage renal disease patients on hemodialysis: a randomized phase 2 trial. Commun Med (Lond). 2024 Jul 26;4(1):153. doi: 10.1038/s43856-024-00575-y. PMID 39060370
- [Derived] Tucker EI, Verbout NG, Markway BD, Wallisch M, Lorentz CU, Hinds MT, Shatzel JJ, Pelc LA, Wood DC, McCarty OJT, Di Cera E, Gruber A. The protein C activator AB002 rapidly interrupts thrombus development in baboons. Blood. 2020 Feb 27;135(9):689-699. doi: 10.1182/blood.2019002771. PMID 31977000

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 53 participants were screened for the study, 13 of which did not meet eligibility criteria. The remaining 40 patients were enrolled. Four participants terminated the study prior to randomization either by withdrawing consent or at the PI's discretion. The remining 36 participants were randomized and dosed on Study Day 1.
Groups:
- AB002 (E-WE-thrombin) Dose 1: Participants received a single dose of 1.5 mcg/kg E-WE thrombin.
  AB002 Dose 1: AB002 (E-WE thrombin) 1.5 mcg/kg administered on Day 1 as a single intravenous infusion
- AB002 (E-WE-thrombin) Dose 2: Participants received a single dose of 3.0 mcg/kg E-WE thrombin.
  AB002 Dose 2: AB002 (E-WE thrombin) 3.0 mcg/kg administered on Day 1 as a single intravenous infusion
- Placebo: Participants received a single dose of placebo
  placebo: placebo administered on Day 1 as a single intravenous infusion
Period: Pre-dose Period (Study Days -7, -5, -2)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Dosing Period (Study Day 1)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Recovery Period (Study Day 3)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Follow-up Period (Study Day 14)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Started | 12 | 12 | 12
Completed | 12 | 11 | 12
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.29) | 53.3 (9.56) | 54.6 (12.3) | 54.2 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 8 | 9 | 9 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 12 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 12 | 33
  White | 1 | 2 | 0 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Treatment-emergent Adverse Events (TEAEs) Related to Treatment Will be Summarized Using Frequency Counts (Safety and Tolerability)
Description: TEAEs will be determined by physical examination that will include assessment of skin, head, ears, eyes, nose, throat, respiratory system, cardiovascular system, gastrointestinal system, neurological condition, blood and lymphatic systems, and the musculoskeletal system.
Time Frame: 22 days
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

2. Primary Outcome: The Number of TEAEs Related to Treatment Will be Summarized Using Frequency Counts (Safety and Tolerability).
Description: as for outcome 1
Time Frame: 22 days
Measure: Number; unit: number of TEAEs related to treatment
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
number of TEAEs related to treatment | 0 | 0 | 0

3. Primary Outcome: The Number of Subjects With Bleeding at the Hemodialysis (HD) Vascular Access Site (Safety and Tolerability)
Description: The number of patients in which clinically relevant and non-major bleeding events occurred from the vascular access site. Bleeding from the access site was assessed immediately following decannulation. Pressure was placed on the access site for 10 min. After 10 minutes, the access site was checked for bleeding. If still bleeding, pressure was applied for another 5 minutes and checked again. This was repeated until hemostasis was achieved and the time to hemostasis was recorded. A time greater than 10 min was considered a non-major bleeding event.
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Population: Two patients from the placebo group had catheters as venous access sites and therefore, time to hemostasis could not be evaluated in these pateints.
Measure: Number; unit: participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 10
participants
  Pre-dose hemodialysis sessions (days -7, -5, -2) | 3 | 2 | 1
  Dosing day hemodialysis session (day 1) | 1 | 0 | 3
  Recovery day hemodialysis session (day 3) | 4 | 0 | 1

4. Primary Outcome: The Number of Subjects With Abnormal Electrocardiogram That is Related to Treatment Will be Summarized Using Frequency Counts (Safety and Tolerability).
Description: 12-lead electrocardiogram measurement. Abnormal electrocardiogram was determined by the study PI. The result was determined to be treatment related if the abnormal electrocardiogram occurred post-treatment and not pre-treatment. Data from the specified time points (Study Day 1 (0.5h post-dose) and Study Day 3) were combined by adding the number of participants on each Study Day that showed an abnormal electrocardiogram compared to pre-treatment (Study Day -8).
Time Frame: Study Days -8 (pre-treatment), Day 1, and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

5. Primary Outcome: The Number of Subjects That Develop Antibodies to Endogenous Thrombin Will be Summarized Using Frequency Counts (Safety and Tolerability).
Description: Immunogenicity measured by the presence of serum anti-thrombin antibodies in both an ADA screening assay and confirmatory assay.
Time Frame: Study day 1 pre-dose and study day 14
Population: Day 14 sample was not collected from one subject in the 3.0 mcg/kg AB002 group.
Measure: Number; unit: participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
participants
  Study day 1 pre-dose | 3 | 5 | 5
  Study day 14: number analyzed (Participants) | 12 | 11 | 12
  Study day 14 | 2 | 3 | 6

6. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Body Temperature in Relation to Treatment Will be Assessed.
Description: Body temperature will be measured in degrees Celsius. Clinically significant changes in body temperature were determined by the study PI. The result was determined to be treatment related if the change in body temperature occurred post-treatment and not pre-treatment. Data from the specified time points (Study Day 1 (1h post-dose) and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in body temperature compared to pre-treatment (Study Days -7, -5, -2, and 1 (pre-dose)).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

7. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Respiratory Rate and Relation to Treatment Will be Assessed.
Description: Respiratory rate will be measured in breaths per minute. Clinically significant changes in respiratory rate were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in respiratory rate occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 (1h post-dose) and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in respiratory rate compared to pre-treatment (Study Days -7. -5. -2 and 1 (pre-dose)).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

8. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Blood Pressure (Systolic and Diastolic) and Relation to Treatment Will be Assessed.
Description: Systolic and diastolic blood pressure will be measured in mmHg. Clinically significant changes in blood pressure were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in blood pressure occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 (1h post-dose) and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in blood pressure compared to pre-treatment (Study Days -7, -5, -2 and 1 (pre-dose)).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 1

9. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Heart Rate and Relation to Treatment Will be Assessed.
Description: Heart rate will be measured in beats per minute. Clinically significant changes in heart rate were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in heart rate occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 (1h post-dose) and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in heart rate compared to pre-treatment (Study Days -7, -5, -2 and 1 (pre-dose)).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

10. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Activated Partial Thromboplastin Time (aPTT) and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Plasma aPTT will be measured in seconds. Clinically significant changes in aPTT were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in aPTT occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in aPTT compared to pre-treatment (Study Days -7, -5, -2 and 1 (pre-dose)).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

11. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Prothrombin Time and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Prothrombin time will be measured in seconds. Clinically significant changes in prothrombin time were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in prothrombin time occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 and Study Day 3) were combined by adding the number of participants on each Study Day that showed a clinically significant change in prothrombin time compared to pre-treatment.
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

12. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Plasma Fibrinogen and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Plasma fibrinogen will be measured in mg/dL. Clinically significant changes in fibrinogen were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in fibrinogen occurred post-treatment compared to pre-treatment. Data from the specified time points (Study Day 1 and Study Day 3, before and after hemodialysis) were combined by adding the number of participants on each Study Day that showed a clinically significant change in fibrinogen compared to pre-treatment (Study Days -7. -5. -2).
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

13. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Thrombin Time and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Thrombin time will be measured in seconds. Clinically significant changes in thrombin time were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in thrombin time occurred post-treatment compared to pre-treatment. Data from the post-treatment time points (Study Day 1 and Study Day 3, before and after hemodialysis) were combined by adding the number of participants on each Study Day that showed a clinically significant change in prothrombin time compared to pre-treatment.
Time Frame: Study days -7, -5, -2 (pre-treatment), 1 and 3 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

14. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Bilirubin (Total and Direct) Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Bilirubin (total and direct) levels in the blood will be measured in mg/dL. Clinically significant changes in bilirubin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in bilirubin occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in bilirubin compared to pre-treatment (Study Day -8).
Time Frame: Study days -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

15. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alkaline Phosphatase Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Alkaline phosphatase levels in the blood will be measured in U/L. Clinically significant changes in alkaline phosphatase were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in alkaline phosphatase occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in alkaline phosphatase compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

16. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Aspartate Aminotransferase (AST) Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: AST levels in the blood will be measured in U/L. Clinically significant changes in aspartate aminotransferase (AST) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in AST occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in AST compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

17. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alanine Aminotransferase (ALT) Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: ALT levels in the blood will be measured in U/L. Clinically significant changes in alanine aminotransferase (ALT) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in ALT occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in ALT compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

18. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Lactate Dehydrogenase (LDH) Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: LDH levels in the blood will be measured in U/L. Clinically significant changes in lactate dehydrogenase (LDH) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in LDH occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in LDH compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

19. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Albumin Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Albumin levels in the blood will be measured in g/dL. Clinically significant changes in albumin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in albumin occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in albumin compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

20. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Sodium Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Sodium levels will be measured in mEq/L. Clinically significant changes in sodium levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in sodium levels occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in sodium levels compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

21. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Potassium Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Potassium levels will be measured in mmol/L. Clinically significant changes in potassium levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in potassium levels occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in potassium levels compared to pre-treatment (Study Day -8).
Time Frame: Study days -8 and 3.
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

22. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Chloride Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Chloride levels will be measured in mEq/L. Clinically significant changes in chloride levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in chloride levels occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in chloride levels compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

23. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Glucose Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Blood glucose levels will be measured in mg/dL. Clinically significant changes in glucose levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in glucose occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in glucose compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

24. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Creatinine Levels and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Creatinine levels will be measured in mg/dL. Clinically significant changes in creatinine levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in creatinine levels occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in creatinine compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

25. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hemoglobin Levels and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hemoglobin levels will be measured in g/dL. Clinically significant changes in hemoglobin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in hemoglobin occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in hemoglobin compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

26. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hematocrit and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hematocrit levels will be measured in %. Clinically significant changes in hematocrit were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in hematocrit occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in hematocrit compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

27. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Total Leukocyte Counts and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Total leukocyte counts will be measured in 10˄3/uL. Clinically significant changes in total leukocyte count were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in total leukocyte count occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in total leukocyte count compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

28. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Differential Leukocyte Counts and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Differential leukocyte counts will be measured in %. Clinically significant changes in differential leukocyte counts were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in differential leukocyte counts occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in differential leukocyte counts compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

29. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Red Blood Cell Count and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Red blood cell count will be measured in 10˄6/uL. Clinically significant changes in red blood cell counts were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in red blood cell counts occurred post-treatment compared to pre-treatment. Data from the post-treatment time point (Study Day 3) is presented as the number of participants that showed a clinically significant change in red blood cell counts compared to pre-treatment (Study Day -8).
Time Frame: Study day -8 and 3
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

30. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Platelet Count and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Platelet count will be measured in 10˄3/uL. Clinically significant changes in platelet count were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in platelet count occurred post-treatment compared to pre-treatment. Data from the post-treatment time points (Study Days 1 and 3) are combined by adding the number of participants on each Study Day that showed a clinically significant change in platelet count post-treatment compared to pre-treatment (Study Days -7, -5, -2).
Time Frame: Study days -7, -5, -2, 1, and 3, pre- and post-dialysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants | 0 | 0 | 0

31. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine pH and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: pH of the urine will be measured.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

32. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Specific Gravity and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Specific gravity of the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

33. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Protein Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Protein levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

34. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Glucose Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Glucose levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

35. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Ketone Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Ketone levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

36. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Bilirubin Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Bilirubin levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

37. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Blood Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Blood levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

38. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Nitrite Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Nitrite levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

39. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Urobilinogen Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Urobilinogen levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

40. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Leukocyte Esterase Levels and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Leukocyte esterase levels in the urine will be evaluated.
Time Frame: Study day -8 and 3
Population: All patients on study were anuric.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Hemodialysis Efficiency as Measured by Frequency of Clotting on the Dialysis Filters and Circuit (Pharmacodynamic Outcome).
Description: Assessment of thrombus accumulation in the dialyzer cartridge measured by visual inspection. Assessment of thrombus accumulation in the dialysis filter measured by visual inspection. A score ranging from 1-6 is determined by someone blinded to treatment by the Visual Score Assessment of Clotting in the Hemodialysis Circuit scale: 1- no clotting/clean dialyzer or few blood streaks affecting less than 5% of the fibers seen at the surface of the dialyzer, 2- blood streaks affecting more than 5% but less than 25% of the fibers seen at the surface of the dialyzer, 3- blood streaks affecting more than 25% but less than 50% of the fibers seen at the surface of the dialyzer, 4- blood streaks affecting more than 50% but less than 75% of the fibers seen at the surface of the dialyzer, 5- blood streaks affecting more than 75% of the fibers seen at the surface of the dialyzer, and 6- complete occlusion, coagulated filter (treatment cannot continue without replacement of dialyzer).
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Measure: Geometric Mean (Standard Error); unit: average visual score of dialyzer filter
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
average visual score of dialyzer filter
  Non-dose days (study days -7, -5, -2, and 3) | 2.58 (0.18) | 2.98 (0.44) | 2.65 (0.25)
  Dose day (study day 1) | 1.50 (0.19) | 2.33 (0.28) | 2.50 (0.29)

42. Secondary Outcome: Hemodialysis Efficiency as Measure by the Frequency of Clotting on the Dialysis Circuit: Venous Chamber (Pharmacodynamic Outcome)
Description: Assessment of thrombus accumulation in the dialysis venous chamber measured by visual inspection. A score ranging from 1-7 is determined by someone blinded to treatment using a Visual Score Assessment of Clotting in the Hemodialysis Circuit: 1- no detectable clotting, 2- presence of fibrous ring or minimum clot affecting less than 5% of chamber space, 3- clot formation, affecting more than 5% but less than 25% of chamber space, 4- clot formation, affecting more than 25% but less than 50% of chamber space, 5- clot formation, affecting more than 50% but less than 75% of chamber space, 6- clot formation, affecting more than 75% of chamber space, and 7- Complete occlusion of chamber.
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Measure: Geometric Mean (Standard Error); unit: average visual score of venous chamber
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
average visual score of venous chamber
  Non-dose days (study days -7, -5, -2, and 3) | 2.99 (0.36) | 3.31 (0.49) | 3.21 (0.38)
  Dose day (study day 1) | 1.25 (1.18) | 1.58 (1.23) | 3.17 (0.61)

43. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Urea Nitrogen (BUN) Levels, URR (Pharmacodynamic Outcome).
Description: Assessment of BUN (mg/dL) before and after hemodialysis as urea reduction ratio (URR), %.
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Population: In some instances, the pre-and post-dialysis values appeared to be switched and were excluded from the summary statistics or a value was missing or not reportable.
Measure: Geometric Mean (Standard Deviation); unit: Urea reduction ratio (%)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Urea reduction ratio (%)
  Pre-dose, day -7: number analyzed (Participants) | 12 | 11 | 11
  Pre-dose, day -7 | 69.48 (5.457) | 68.16 (6.419) | 69.68 (6.172)
  Pre-dose, day -5: number analyzed (Participants) | 11 | 12 | 7
  Pre-dose, day -5 | 70.48 (5.709) | 68.43 (6.646) | 71.44 (6.975)
  Pre-dose, day -2: number analyzed (Participants) | 10 | 10 | 11
  Pre-dose, day -2 | 68.51 (7.467) | 68.62 (6.496) | 68.69 (6.849)
  Post-dose, day 1: number analyzed (Participants) | 12 | 11 | 11
  Post-dose, day 1 | 70.63 (6.955) | 70.61 (5.146) | 69.77 (6.135)
  Post-dose (recovery), day 3: number analyzed (Participants) | 10 | 12 | 12
  Post-dose (recovery), day 3 | 69.09 (7.599) | 69.21 (6.391) | 67.08 (8.132)

44. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Urea Nitrogen (BUN) Levels (Pharmacodynamic Outcome), KtV.
Description: Assessment of BUN (mg/dL) before and after hemodialysis as KtV (mL/min).
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Population: as for outcome 43
Measure: Geometric Mean (Standard Deviation); unit: KtV (mL/min)
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
KtV (mL/min)
  Pre-dose day -7: number analyzed (Participants) | 12 | 11 | 11
  Pre-dose day -7 | 1.411 (0.2261) | 1.367 (0.2597) | 1.392 (0.2505)
  Pre-dose day -5: number analyzed (Participants) | 11 | 12 | 7
  Pre-dose day -5 | 1.436 (0.2025) | 1.343 (0.2429) | 1.470 (0.2408)
  Pre-dose day -2: number analyzed (Participants) | 10 | 10 | 11
  Pre-dose day -2 | 1.372 (0.2657) | 1.391 (0.2427) | 1.388 (0.2357)
  Post-dose day 1: number analyzed (Participants) | 12 | 11 | 11
  Post-dose day 1 | 1.468 (0.2542) | 1.553 (0.4112) | 1.418 (0.2312)
  Post-dose day 3: number analyzed (Participants) | 10 | 12 | 12
  Post-dose day 3 | 1.381 (0.2437) | 1.373 (0.2366) | 1.319 (0.2908)

45. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Potassium Levels (Pharmacodynamic Outcome).
Description: Assessment of plasma potassium (mmol/L) before and after hemodialysis. The reduction of plasma potassium is reported as fold change (post-hemodialysis plasma potassium/ pre-hemodialysis plasma potassium).
Time Frame: At each hemodialysis session (non-dose days: study day -7, -5, -2, and 3 and dose day: study day 1)
Population: In some instances, the pre-and/or post-dialysis values appeared to be switched and were excluded from the summary statistics or a value was missing or not reportable.
Measure: Geometric Mean (Standard Deviation); unit: fold change plasma potassium
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
fold change plasma potassium
  Pre-dose day -7: number analyzed (Participants) | 12 | 11 | 11
  Pre-dose day -7 | 0.78 (0.066) | 0.75 (0.091) | 0.71 (0.064)
  Pre-dose day -5: number analyzed (Participants) | 11 | 12 | 8
  Pre-dose day -5 | 0.72 (0.068) | 0.83 (0.337) | 0.70 (0.068)
  Pre-dose day -2: number analyzed (Participants) | 11 | 11 | 11
  Pre-dose day -2 | 0.75 (0.076) | 0.73 (0.116) | 0.70 (0.099)
  Post-dose day 1: number analyzed (Participants) | 12 | 11 | 11
  Post-dose day 1 | 0.73 (0.074) | 0.75 (0.16) | 0.68 (0.085)
  Post-dose day 3: number analyzed (Participants) | 11 | 12 | 12
  Post-dose day 3 | 0.72 (0.083) | 0.76 (0.07) | 0.75 (0.087)

46. Secondary Outcome: The Effect of a Single Intravenous Dose of E-WE Thrombin on Plasma Activated Protein C-Protein C Inhibitor Complex (APC-PCI) Levels as a Surrogate for Drug Exposure.
Description: Plasma APC-PCI (ng/mL) levels will be determined by ELISA.
Time Frame: Study day 1: (pre-dose, 0.167h, 0.5h, 1h, 2h, 4h, 6h, 24h post-dose)
Population: In some samples the values were missing or not reportable.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
ng/mL
  pre-dose | 0.1808 (0.6264) | 1.447 (1.749) | 0.9508 (1.885)
  0.167h: number analyzed (Participants) | 12 | 12 | 10
  0.167h | 31.03 (8.300) | 54.29 (18.67) | 0.2480 (0.7842)
  0.5h: number analyzed (Participants) | 12 | 12 | 10
  0.5h | 54.00 (21.03) | 97.01 (31.41) | 0.4310 (1.363)
  1h | 62.52 (24.50) | 103.9 (37.62) | 0.7736 (1.842)
  2h: number analyzed (Participants) | 12 | 12 | 11
  2h | 57.77 (25.31) | 95.92 (36.50) | 2.441 (3.780)
  4h | 58.52 (26.79) | 80.38 (33.06) | 6.094 (5.036)
  6h: number analyzed (Participants) | 11 | 12 | 7
  6h | 11.33 (7.265) | 13.80 (5.383) | 2.740 (2.168)
  24h: number analyzed (Participants) | 12 | 12 | 5
  24h | 0.2808 (0.9728) | 0.4067 (0.9562) | 1.962 (2.034)

47. Secondary Outcome: The Number of Subjects That Develop Anti-drug Antibodies Will be Summarized by Frequency Counts.
Description: Plasma anti-drug antibodies will be determined by ELISA.
Time Frame: Study day 1 pre-dose and study day 14
Population: Day 14 sample was not collected from one participant in the 3.0 mcg/kg AB002 group.
Measure: Count of Participants; unit: Participants
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Study day 1 pre-dose | 0 | 1 | 1
  Study day 14 post-dose: number analyzed (Participants) | 12 | 11 | 12
  Study day 14 post-dose | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study check-in (Day -8) through the final follow-up (Day 14) for a total of 22 days.
Arm/Group | AB002 (E-WE-thrombin) Dose 1 | AB002 (E-WE-thrombin) Dose 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB002 (E-WE-thrombin) Dose 1 (N=12) | AB002 (E-WE-thrombin) Dose 2 (N=12) | Placebo (N=12)
baclofen toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB002 (E-WE-thrombin) Dose 1 (N=12) | AB002 (E-WE-thrombin) Dose 2 (N=12) | Placebo (N=12)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Aronora, Inc. shall retain title to and the right to publish all documentation, records, raw data, specimens, or other work product generated in connection with this study. Such publications shall not be made by the PI or Celerion without the prior written consent of Aronora, Inc.

DOCUMENTS (3):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03963895/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03963895/SAP_001.pdf
  • Informed Consent Form (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT03963895/ICF_002.pdf